CLINICAL TRIAL: NCT00569088
Title: "973" Project for Pathology of Traditional Chinese Medicine
Brief Title: Study of the Pathogenesis and Molecular Mechanism of "YURE" in Internal Intractable Diseases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Mianhua Wu, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006CB504807
Record Dates: First submitted 2007-11-28; First posted 2007-12-06 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Stroke
Keywords: hemorrhagic stroke; Chinese Medicine; pathogenesis; YURE
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): A combined treatment would be used in the arm.That means Chinese herb formula would be used with the current Modern Medicine therapy for stroke in this arm.
  Interventions: Drug: Chinese herbs formula
- A (Active Comparator): just the current Modern Medicine therapy for stroke would be available in the arm.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Chinese herbs formula — The chinese herbs formula includes eight herbs,and they are Radix et Rhizoma Rhei Palmati(Rhubarb,10 grams),Cornu Bubali(Buffalo Horn,30 grams),Radix Paeoniae Bubra(Red Peony Root,15 grams),Cortex Moutan Radicis(Tree Peony Root-bark,10 grams),Radix Rehmanniae(Adhesive Rehmannia Root Tuber,20 grams),Pheretima Aspergillum(Earth-worm,10 grams),Radix Notoginseng(Sanchi,5 grams)and Rhizoma Acori Tarainowii(Tararinow Sweetflag Rhizome,10 grams).
  Boiled together. 150ml of the juice,p.o.,twice a day,for 28 days
  Arms: B
Drug: Mannitol — 250 ml Mannitol Injection or Glycerin and Fructose Injection ,once a day, for 3-5 days
  Arms: A

SUMMARY:
The purpose of this study is to determine whether the Chinese herbs formula is effective in the treatment of hemorrhagic stroke and to find out Chinese pathogeny and pathogenesis in the disease.

DETAILED DESCRIPTION:
Blood stasis and blood heat are two pathogens in the theory system of Chinese Medicine, which can cause many diseases independently. But in internal intractable diseases, such as viral hepatitis, stroke, and epidemic hemorrhagic fever, blood stasis and blood heat always accompany with each other. So the hypothesis is raised that blood stasis with heat (YURE) is a compound pathogen and key pathogenesis in internal intractable diseases. This study was aimed to verify the role that the compound pathogen played in hemorrhagic stroke and to observe the progress of the key pathogenesis. A randomized and controlled trial would be conducted in five hospitals, where 300 hospitalized patients with hemorrhagic stroke in the acute phase would receive different intervention with basic modern medicine treatment or Chinese herbs formula combined with the former. The Chinese herbs formula, which was designed under the guidance of the theory system of Chinese Medicine, was supposed to cool blood heat and dissolve blood stasis. Clinical efficacy and safety would be evaluated after the 21-days intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hemorrhagic stroke
* hospitalized in 48 hours after hemorrhagic stroke happens

Exclusion Criteria:

* Subarachnoid Hemorrhage
* intracranial hemorrhage caused by tumor, trauma or blood diseases

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Chinese symptoms | 21 days

SECONDARY OUTCOMES:
blood loss determined by brain CT | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Mianhua Wu, Dr., Principal Investigator — Nanjing Uinversity of Traditional Chinese Medicine
Locations (1):
- Institute of Internal Intractable Diseases, Nanjing University of Traditonal Chinese Medicine, Nanjing, Jiangsu, China